CLINICAL TRIAL: NCT02178085
Title: Ocular Blood-flow Assessment by Magnetic Resonance Angiography in Glaucoma
Brief Title: Ocular Blood Flow Assessment in Glaucoma
Acronym: OBAMAg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2014_843_0007; 2014-A00847-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-06-18; First posted 2014-06-30 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Glaucoma
Keywords: glaucoma; phase-contrast MRI; blood flow; cerebrospinal fluid
MeSH Terms: conditions — Glaucoma | interventions — Cerebrovascular Circulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flow imaging (Experimental): Glaucoma patients and healthy subjects who will undergo ocular flow imaging
  Interventions: Other: Flow imaging

INTERVENTIONS:
Other: Flow imaging — Participants will undergo morphological and then flow MRI. Flow MR images will be processed adequately to obtain quantitative values of arterial and venous flow as well as CSF flow.
  Other Names: Flow MRI; Cine phase-constrast magnetic resonance imaging; Cerebral blood flow

SUMMARY:
Background : Glaucoma is a common disease, potentially blinding, characterized by progressive damage to the optic nerve. If the intraocular pressure is the most known risk factor, however, there are cases of glaucoma scalable despite well-controlled intraocular pressure, ocular hypertension without glaucoma or glaucoma without ocular hypertension (normal tension glaucoma).

Purpose :Involvement of vascular factors in the development of glaucoma and scalability has been proved, associated with a possible loss of vascular autoregulation. The objective of this study is to quantify MRI flow of blood flows referred ophthalmic patients with glaucoma untreated comparison with control subjects.

DETAILED DESCRIPTION:
Eye vascularization, supplied by ophthalmic artery and superior ophthalmic vein is not easily accessible to routine explorations to date. Similarly the potential oscillations of the cerebrospinal fluid (CSF) around the optic nerve have not been described. Developments in magnetic resonance imaging (MRI) provide new insights into the quantitative study of blood and CSF flows through phase contrast MRI also called "flow MRI". Our hypothesis is that the ability of MRI to measure intracranial flow is applicable to the vasculature of the eye.

The MRI protocol will be applied to control adult subjects previously examined by an ophthalmologist. Structures to be imaged will be identified on a morphological sequence. Each MRI phase contrast slice (flow MRI) will be positioned perpendicularly to the flow direction. The flow MRI data will be analysed by a dedicated image processing tool which performs the vessels segmentation. For each curve of the vessel flow evolution during the cardiac cycle is reconstructed.

Glaucomatous patients will undergo a six-month follow-up to determine if they respond to their therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants
* Diagnosis of primary open angle glaucoma or normal-tension glaucoma
* Never received any anti glaucoma therapy
* Patients included in the group " normal pressure glaucoma " are patients where the diagnosis of optic neuropathy have been worn by the ophthalmologist with measured intraocular pressure <21 mmHg.
* Healthy controls will be examined by an ophthalmologist before inclusion

Exclusion Criteria:

* Anyone with a classic contraindication to MRI
* Cardiovascular comorbidities or neurovascular : uncontrolled systemic hypertension , Diabetes, heart failure , carotid stenosis , ischemic stroke or transient ischemic attack.
* Already treated glaucoma
* Prescription by the ophthalmologist another treatment than prostaglandin analogue treatment.
* Other clinical forms of glaucoma : angle closure glaucoma, neovascular glaucoma, exfoliative glaucoma, secondary glaucomas, pigment dispersion glaucoma, traumatic glaucoma, congenital glaucoma
* Presence of other ocular pathology (simple refractive error allowing 10/10 of best corrected visual acuity and mild and moderate cataracts will not be considered as a criterion for non- inclusion).
* History of intraocular or orbital surgery of less than 6 months .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Arterial blood flow | Day 1
  Measure of the mean arterial blood flow during the cardiac cycle in the ophthalmic artery.

SECONDARY OUTCOMES:
Vascular flow curves | Day 1
  Temporal and amplitude parameters of vascular flow curves (arteries and veins)
Cerebrospinal fluid (CSF) dynamic | Day 1
  Temporal and amplitude parameters of cerebrospinal fluid (CSF) curves measured in the optic nerve sheath.
Treatment response | Day 180
  Determination of treatment response
  1. Measurement of ocular tone (21 mmHg threshold under which the patient may be responder to treatment value)
  2. Extent of the visual field (if stable patient responder)
  3. Measure optic disc (if stable patient responder)
  The three conditions must be true to declare a patient responder to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Balédent, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens, Amiens, Picardie
  - Centre d'ophtalmologie Victor Pauchet, Amiens, Picardie